CLINICAL TRIAL: NCT02139072
Title: Accuracy of CoaguChek XS in Patients With Antiphospholipid Antibody Syndrome
Brief Title: CoaguChek XS in Antiphospholipid Antibody Syndrome (APL) Patients
Status: Completed | Type: Observational
Sponsor: University of Florida (Other)
Collaborators: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Other Study IDs: IRB201400096
Record Dates: First submitted 2014-05-13; First posted 2014-05-15 (Estimated); Last update posted 2016-10-04 (Estimated); Status verified 2016-01

CONDITIONS: Antiphospholipid Antibody Syndrome
Keywords: Anticoagulation; International normalized ratio; Warfarin
MeSH Terms: conditions — Antiphospholipid Syndrome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- CoaguChek XS: INR measured by CoaguChek XS in patients with APL at visit 1 and visit 2, in addition to routine measure by standard lab draw
  Interventions: Device: CoaguChek XS; Procedure: Standard Lab Draw
- Standard Lab Draw: INR measured by standard lab draw at visit 1 and visit 2 for non-APL patients, in addition to routine measurement by CoaguChek XS
  Interventions: Device: CoaguChek XS; Procedure: Standard Lab Draw

INTERVENTIONS:
Device: CoaguChek XS — CoaguChek XS will be used to measure INR in patients with APL
Procedure: Standard Lab Draw — Patients on warfarin for any indication other than APL will measure INR by venous lab draw

SUMMARY:
The purpose of this study is to see if the CoaguChek XS is accurate in measuring International Normalized Ratio (INR) in patients with Antiphospholipid Antibody Syndrome (APL) receiving warfarin therapy.

DETAILED DESCRIPTION:
Antiphospholipid Antibody Syndrome (APL) is an autoimmune disease that increases ones risk for blood clots. Therefore, these patients receive anticoagulation therapy with warfarin. Point of care devices such as the CoaguChek XS are often used to monitor International Normalized Ratio (INR) in patients on warfarin. However, the antibodies present in patients with APL may lead to false INR results when using the CoaguChek XS. This study will compare the accuracy of the CoaguChek XS in measuring INR in patients with APL by measuring INR by the CoaguChek XS and a standard lab as a reference point. Patients on warfarin for indications other than APL will be measured by both methods as well to serve as a control group.

ELIGIBILITY:
Inclusion Criteria:

* 18-65 years of age
* anticoagulated with warfarin for at least 1 month
* Diagnosis of antiphospholipid antibody syndrome for intervention arm

Exclusion Criteria:

* any type of mental disability that would hinder their ability to give informed consent
* any terminal illness or any other condition that could interfere with study completion, that person will be excluded.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients presenting to UF/Shands Hematology Anticoagulation Clinic for a routine office visit with pharmacy.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2015-03; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
International Normalized Ratio (INR) | Day 1 and Day 60
  Compare INR obtained by CoaguChek XS to INR obtained from venous lab draw. Difference of +/- 0.5 considered significant

CONTACTS AND LOCATIONS:
Overall Officials: James Taylor, PharmD, Principal Investigator — University of Florida
Locations (1):
- UF and Shands Health, Gainesville, Florida, United States